CLINICAL TRIAL: NCT01617915
Title: Tumor Specific Plasma DNA
Status: Completed | Type: Observational
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Gary Schwartz, Associate Professor of Medicine, Dartmouth-Hitchcock Medical Center
Other Study IDs: D12127
Record Dates: First submitted 2012-06-10; First posted 2012-06-13 (Estimated); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Breast Cancer; Lung Cancer
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
In 2011, there was an estimated 233,000 cases of invasive breast cancer, and 39,970 deaths from breast cancer in the United States. The vast majority of patients are diagnosed with Stage I-III resectable and potentially curable disease, and for these patients, the most pressing questions are whether adjuvant endocrine or chemotherapy are indicated, and if so, how to determine whether these treatments are working. Adjuvant systemic therapy reduces relative recurrence rates by 30-50%, depending on the age of the patient and tumor characteristics. However, patients with early stage disease often do not bear measurable markers of disease such as an elevated cancer antigen 27-29 (CA27.29) or circulating tumor cells. Patients with early stage breast cancer are typically treated with adjuvant therapy based on historical evidence showing that such therapy prolongs survival in this population.

Lung cancer is the most common malignancy and the leading cause of cancer-related death in the U.S. Approximately 220,000 new cases of lung cancer are diagnosed in the U.S. every year. Unfortunately, lung cancers are often diagnosed at later stages than breast cancer, due in part to little/no effective screening for lung cancer. As with breast cancer, patients are commonly treated with chemotherapeutic agents, but treatment regimens can take several weeks to months to elicit clinically detectable anti-tumor effects. A biomarker to assess early tumor response to therapy would benefit this patient population.

The contents of dying tumor cells can be detected in the bloodstream, and this may be enhanced by the leaky vasculature of solid tumors. Protein biomarkers of tumor cell death are difficult to detect due to the complex nature of plasma and the lack of technical sensitivity. In contrast, DNA is easier to detect through polymerase chain reaction (PCR) amplification. Indeed, circulating tumor DNA has been detected in plasma from patients with osteosarcoma, breast cancer, and colorectal cancer. Until recently, it was impractical to develop an assay to routinely quantify circulating tumor DNA due to heterogeneity between patients and tumors. Advances in genomic technology now permit sequencing a tumor genome to identify patient-specific genomic aberrations. Major genomic alterations (i.e., insertions, amplifications, deletions, inversions, translocations) can be readily detected using PCR primers which will recognize tumor DNA but not normal DNA.

While this strategy may be generally applicable to diverse types of solid tumors, two issues are apparent in breast cancer. Firstly, the incidence of chromosomal rearrangements varies widely. Whole-genome sequencing of 15 breast tumors revealed a range of 1-231 major genomic alterations (mean= 68), where 2 tumors had 1 alteration, and 9 tumors had > 20 alterations. Single-base point mutations are more common but difficult to reliably detect using PCR. Therefore, the investigators must consider that a small subset of patients may have a limited number of genomic alterations available for this assay. Secondly, intratumoral heterogeneity may mean that some genomic alterations are not present in every tumor cell. Such heterogeneity has been inferred from FISH and immunohistochemistry (IHC) studies for many years, and is now being verified at the genomic level. The investigators must consider that only a subpopulation of tumor cells may be sensitive to cytotoxic therapy, so changes in the levels of circulating tumor DNA may only be reflected with analysis of genomic alterations specific to the sensitive cells.

ELIGIBILITY:
Inclusion Criteria:

Women or men > age 18.

Ability to give informed consent

Archived tumor tissue must be available for genetic analysis.

Patients with early-stage breast cancer

Histologic documentation of invasive breast cancer by core needle or incisional biopsy.

The invasive cancer must be either:

* triple-negative with both estrogen and progesterone receptor staining present in fewer than 10% of invasive cancer cells by IHC, and HER2-negative defined as IHC 0-1+, or with a FISH ratio of <1.8 if IHC is 2+ or if IHC has not been done.

or

*HER2-positive with IHC 3+ or a FISH ratio of >2.2.

Clinical Stage II-III invasive breast cancer with the intent to treat with:

* pretreatment mammography, ultrasound, and breast MRI for staging
* pretreatment axillary staging
* neoadjuvant treatment with DNA-damaging chemotherapy (with or without HER2- directed therapy)
* post-chemotherapy breast MRI
* surgical resection of the primary tumor with an axillary dissection for one or more positive nodes after neoadjuvant chemotherapy

Patients with multicentric or bilateral disease are eligible if the target lesion(s) meet the other eligibility criteria.

No prior chemotherapy, endocrine therapy, or radiotherapy with therapeutic intent for treatment of a prior malignancy is allowed.

Patients with locally advanced or metastatic breast cancer Histologic documentation or history of invasive breast cancer by core needle or incisional biopsy, or by surgical resection.

ER/PR/HER2 status may be determined using any breast tumor specimen acquired at any point during a given patient's disease history (i.e., archived tumor). The invasive cancer must be either:

*triple-negative with both estrogen and progesterone receptor staining present in fewer than 10% of invasive cancer cells by IHC, and HER2-negative defined as IHC 0-1+, or with a FISH ratio of <1.8 if IHC is 2+ or if IHC has not been done.

or

*HER2-positive with IHC 3+ or a FISH ratio of >2.2.

Clinical Stage III-IV invasive breast cancer not amenable to curative surgical resection, with intent to treat with:

* if tumor is triple-negative, treatment with DNA-damaging chemotherapy as per standard of care in the first-line setting for advanced/metastatic disease.
* if tumor is HER2+, treatment with DNA-damaging chemotherapy, HER2-directed therapy, or a combination as per standard of care in any setting for advanced/metastatic disease.
* CT of chest, abdomen, and pelvis and bone scan or PET-CT for staging to assess response (by RECIST) approximately every 8 weeks or as clinically indicated with the primary course of DNA-damaging chemotherapy. The bone scan will not need to be repeated if the baseline bone scan is negative.

Patients with newly diagnosed non-small cell lung cancer (NSCLC) Histologic documentation of NSCLC by core needle biopsy or a fine needle aspirate.

Clinical Stage II or III lung cancer with the intent to treat with:

* pretreatment chest CT and or PET/CT
* induction (neoadjuvant) therapy with DNA-damaging chemotherapy
* post-chemotherapy lung chest CT and or PET/CT
* surgical resection of the primary tumor(s) after induction (neoadjuvant) chemotherapy No prior chemotherapy or radiotherapy with therapeutic intent for treatment of a prior malignancy is allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast and Lung cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2012-10; Primary Completion 2021-05-07 (Actual); Study Completion 2021-05-07 (Actual)

PRIMARY OUTCOMES:
Circulating tumor levels correlation to response | 6 months
  To determine whether acute increases in the levels of circulating tumor DNA correlate with response to chemotherapy in patients with breast cancer.

SECONDARY OUTCOMES:
Circulating tumor DNA following surgery | 6 months
  To determine whether the levels of circulating tumor DNA acutely decrease following surgical resection of a primary breast tumor.
To determine optimal timing for detection of circulating tumor DNA | 6 months
  To determine the optimal timing for detection of changes in levels of circulating tumor DNA.
Circulating tumor DNA detection following surgery | 6 months
  To determine whether circulating tumor DNA detectable at 1-2 weeks following surgical resection of a primary tumor predicts disease recurrence.
Circulating tumor DNA correlation with pathologic complete response | 6 months
  To determine whether the fall in circulating tumor DNA correlates with pathologic complete response to neoadjuvant chemotherapy in patients with early-stage breast cancer, or with clinical response to chemotherapy in patients with locally advanced or metastatic breast cancer..
Circulating tumor DNA correlation with clinical evidence of disease recurrence or progression | 6 months
  To determine whether circulating tumor DNA levels increase prior to clinical evidence of disease recurrence or progression.

CONTACTS AND LOCATIONS:
Overall Officials: Gary N Schwartz, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States